CLINICAL TRIAL: NCT02630550
Title: Validation of the Cheetah NICOM by Comparison to TEE During Open Vascular Surgery - Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Louis-Philippe Fortier, Department Head - Anesthesia, Maisonneuve-Rosemont Hospital
Other Study IDs: 15042
Record Dates: First submitted 2015-12-02; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Aortic Aneurysm; Peripheral Arterial Disease
Keywords: Cardiac output; Intraoperative Monitoring; Echocardiography, Transesophageal; Vascular cross-clamping; Endarterectomy; Monitoring, Physiologic/instrumentation; Cardiography, Impedance
MeSH Terms: conditions — Aortic Aneurysm; Peripheral Arterial Disease | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Aortic Aneurysm Repair: The impact of large abdominal retractors and an abdominal aortic cross-clamp on the validity of the Cheetah NICOM's measurements will be evaluated in this group.
  Interventions: Device: Cheetah NICOM; Device: Transesophageal echocardiography (TEE)
- Femoral Endarterectomy: The impact of the clamping of a large peripheral arterial vessel on the validity of the Cheetah NICOM's measurements will be evaluated in this group.
  Interventions: Device: Cheetah NICOM; Device: Transesophageal echocardiography (TEE)

INTERVENTIONS:
Device: Cheetah NICOM — The Cheetah NICOM will be installed on all patients to evaluate the validity of its measurements.
Device: Transesophageal echocardiography (TEE) — TEE will serve as gold standard measurements for the evaluation of the Cheetah NICOM.

SUMMARY:
The Cheetah NICOM is a non-invasive cardiac output monitor that has been validated in various clinical contexts but not during the occlusion of major arteries, as takes place in vascular surgery. The present study will evaluate the precision and validity of the measures taken by the device during open vascular surgery procedures. The measurements will be compared to the those calculated by transesophageal echocardiography at various key points during the surgeries. The validity of the cardiac output, stroke volume and stroke volume variation measurements will be evaluated, as well as the device's ability to track rapid changes in cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing an elective open aortic aneurysm repair surgery or a femoral endarterectomy under general anesthesia.
* ASA 1-3

Exclusion Criteria:

* Refuses general anesthesia
* Contraindication to transesophageal echocardiography
* Allergy to the glue of the Cheetah NICOM probes
* Severe aortic valve regurgitation
* Thoracic aorta anatomy anomaly
* Unipolar pacemaker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing either an open aortic aneurysm repair surgery or a femoral endarterectomy under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Validity of Stroke Volume (SV) Measurements by the Cheetah NICOM | Per vascular surgery procedure
  The SV measured by the Cheetah NICOM will be compared to the one measured by transesophageal echocardiography at multiple time points during the surgery.

SECONDARY OUTCOMES:
Stroke Volume (SV) with a vascular cross-clamp | Per vascular surgery procedure when a cross-clamp is installed
  The SV measured by the Cheetah NICOM will be compared to the one measured by transesophageal echocardiography at multiple points once a vascular cross-clamp is installed.
Stroke Volume (SV) trending ability | Per vascular surgery procedure
  Between each pair of consecutive data points, the change of SV measurements given by the Cheetah NICOM will be compared to those given by transesophageal echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Fortier, MD, MSc, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada